CLINICAL TRIAL: NCT06882863
Title: Reducing Sedentary Behavior in Patients with Severe COPD: a Nurse-Led Motivational Intervention
Brief Title: Reducing Sedentary Behavior in Patients with Severe COPD: a Feasibility Study on Nurse-Led Motivational Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SJ-1089
Record Dates: First submitted 2025-03-11; First posted 2025-03-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility (Experimental): This feasibility study involves a single-arm intervention where patients with severe COPD receive nurse-led motivational interviews to reduce sedentary behavior. Participants recieve one 60 minute intervention, focusing on identifying barriers, setting small activity goals, and building motivation using motivational interviewing (MI) and Cognitive Behavioral Therapy (CBT) techniques.
  Participants wear accelerometers for seven days before the intervention to measure changes in sedentary time. The study assesses recruitment feasibility, adherence, and patient acceptability, informing refinements before a future randomized controlled trial (RCT).
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — This intervention consists of a single nurse-led motivational interview aimed at reducing sedentary behavior in patients with severe COPD. The session, conducted in the patient's home, lasts approximately 60 minutes and focuses on identifying personal barriers, exploring motivation, and setting small, realistic goals to reduce sedentary time.
  Unlike traditional pulmonary rehabilitation, this intervention does not involve structured exercise but instead uses motivational interviewing (MI) techniques to encourage gradual behavior change in daily routines. Before the intervention, patients wear an accelerometer for seven days to objectively measure baseline sedentary time. The study assesses feasibility, patient engagement, and adherence to determine whether the approach is suitable for a larger randomized controlled trial (RCT).

SUMMARY:
This feasibility study aims to assess the practicality and acceptability of a nurse-led motivational interview intervention designed to reduce sedentary behavior in patients with severe Chronic Obstructive Pulmonary Disease (COPD). The study will evaluate the recruitment process, patient adherence, and the usability of accelerometers for objectively measuring sedentary time.

A total of 10-12 patients with severe COPD will be recruited and receive individual motivational interviews conducted by trained nurses in their homes. The intervention will be based on motivational interviewing (MI) and Cognitive Behavioral Therapy (CBT) principles, focusing on helping patients identify barriers and set realistic goals to increase physical activity.

The study will determine whether patients tolerate wearing accelerometers for seven days at different time points and whether the intervention is acceptable to both patients and nurses. Insights gained from this feasibility study will guide refinements to the intervention before launching a randomized controlled trial (RCT) to test its effectiveness on a larger scale.

DETAILED DESCRIPTION:
This feasibility study is designed to assess whether a nurse-led motivational interview intervention can be effectively implemented to reduce sedentary behavior in patients with severe Chronic Obstructive Pulmonary Disease (COPD). Severe COPD is associated with breathlessness and functional limitations, which often lead to prolonged sedentary time, increasing the risk of disease progression and reduced quality of life. Although pulmonary rehabilitation programs exist, many patients struggle with participation due to physical discomfort, lack of motivation, or fear of exacerbating their symptoms. This study aims to evaluate whether an intervention focusing on behavioral change and motivation can help patients engage in small but meaningful reductions in sedentary time.

The feasibility study will recruit 10 patients with severe COPD from pulmonary outpatient clinics. Each participant will receive two to three motivational interviews conducted by a trained nurse in their home over a period of three months. The intervention is based on motivational interviewing (MI) and Cognitive Behavioral Therapy (CBT) principles, both of which have shown effectiveness in supporting behavior change. During these sessions, the nurse will help the patient identify their current level of sedentary behavior, explore their personal motivations for change, and work together to develop achievable, realistic strategies to increase physical activity in daily life. The intervention will focus on small, individualized goals, such as standing up during television commercials, incorporating brief walks, or engaging in light household activities, with the aim of making these changes sustainable.

A critical aspect of the study is assessing whether patients are willing and able to wear accelerometers to measure their sedentary time objectively. Each participant will wear an accelerometer for seven consecutive days before the intervention, allowing researchers to evaluate whether the device is tolerated and whether it provides reliable data on activity levels. In addition to the accelerometer data, participants will provide feedback on their experience with the intervention, including how easy or difficult it was to implement suggested changes, whether they found the motivational interviews helpful, and whether they encountered any barriers. Nurses delivering the intervention will also provide feedback on the practicality of the sessions, the level of patient engagement, and any modifications that may be needed to improve the intervention before scaling up to a larger trial.

The study will also examine how well patients adhere to the intervention, tracking how many complete all scheduled sessions and whether they report making changes to their daily activity patterns. By evaluating recruitment success, adherence rates, patient satisfaction, and the usability of accelerometer-based measurements, the study will identify whether the intervention is feasible and acceptable for both patients and healthcare providers. If challenges arise, adjustments will be made to refine the recruitment process, session structure, or measurement methods before proceeding to a full randomized controlled trial (RCT).

The findings from this feasibility study will be used to optimize the intervention and study design, ensuring that a future large-scale trial can be conducted smoothly and effectively. If successful, this nurse-led motivational interview approach could become a valuable component of COPD care, helping patients make meaningful, sustainable reductions in sedentary behavior, improving their overall health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe COPD confirmed by a healthcare provider.
* Aged 65 years or older at the time of enrollment.
* Self-reported sedentary behavior of at least 5 hours per day.
* Able to provide informed consent and participate in a home-based interview.
* Not currently enrolled in a structured pulmonary rehabilitation program.

Exclusion Criteria:

* Severe cognitive impairment that prevents meaningful participation in the motivational interview.
* Physical disability that completely prevents movement and makes physical activity recommendations irrelevant.
* Severe comorbidities with a life expectancy of less than six months.
* Inability to understand or communicate in Danish.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the intervention | From enrollment to one week post-intervention
  Measured by the number of participants who successfully complete the intervention.

SECONDARY OUTCOMES:
questionnaire | From enrollment to one week post-intervention
  Measured by the number of participants who successfully complete the provided questionnaire SF-12
questionnaire | From enrollment to one week post-intervention
  Measured by the number of participants who successfully complete the provided questionnaire CRQ
questionnaire | From enrollment to one week post-intervention
  Measured by the number of participants who successfully complete the provided questionnaire HADS.

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark